CLINICAL TRIAL: NCT05831579
Title: A Phase I Trial of Palliative Spatially Fractionated (GRID) Radiotherapy Using Intensity Modulated Proton Therapy
Brief Title: Palliative Spatially Fractionated (GRID) Radiotherapy Using Intensity Modulated Proton Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202304011
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Unresectable Solid Tumor; Metastatic Cancer
Keywords: proton; palliative radiotherapy; spatially fractionated radiotherapy; GRID; stereotactic body radiotherapy (SBRT); stereotactic ablative radiotherapy (SABR); cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort A: Reirradiation of Treatment Fields (Experimental): Radiotherapy will consist of 20 Gy proton GRID radiotherapy x 3 fractions.
  Interventions: Radiation: Proton GRID Radiotherapy
- Cohort B: De Novo Radiation Treatment Fields (Experimental): Radiotherapy will consist of 20 Gy proton GRID radiotherapy x 3 fractions.
  Interventions: Radiation: Proton GRID Radiotherapy

INTERVENTIONS:
Radiation: Proton GRID Radiotherapy — The proton GRID radiotherapy prescription dose is 20 Gy x 3 fractions to the tumor, with an integrated dose of 6 Gy x 3 fractions to the PTV. Treatment to multiple lesions within the PTV is allowed (ex. a dominant lesion plus satellites). Multiple proton GRID radiotherapy plans may be delivered on the same day or different days, but they cannot overlap.

SUMMARY:
Spatially fractionated radiotherapy (SFRT or GRID) addresses some limitations of traditional stereotactic body radiation therapy by relying on beam collimation to create high-dose "peaks" and intervening low-dose "valleys" throughout the target volume. Standard palliative radiotherapy regimens provide limited durability of response, and there are challenges with delivery to large tumors or in previously irradiated fields. In this study, Proton GRID radiotherapy will be used to deliver three-fraction palliative radiotherapy to patients with tumors needing palliative radiation. The safety and efficacy of this approach will be assessed. It is hypothesized that GRID is highly effective, immunogenic, and associated with low rates of toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cancer diagnosis.
* Planning to undergo palliative radiotherapy to unresectable or metastatic target lesion ≥ 4.5 cm in any dimension as measured with radiographic imaging or with calipers by clinical exam.

  * Cohort A: 10 patients with lesions that have been previously irradiated.
  * Cohort B: 10 patients with lesions that have not been previously irradiated.
* ECOG performance status ≤ 3
* At least 18 years of age.
* Radiotherapy is known to be teratogenic. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 6 months after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Patients with tumors in need of urgent surgical intervention, such as life-threatening bleeding or those at high risk for pathologic fracture and amenable to surgical intervention.
* Patients with a superficial target lesion ≤ 1 cm deep to skin surface who initially had a superficial lesion irradiated, if the target lesion was in the area of the prior irradiation.
* Currently receiving any cytotoxic cancer therapy regimens or VEGF inhibitors that will overlap with the proton GRID administration.
* Cytotoxic chemotherapy and VEGF inhibitors prior to radiotherapy or planned after radiotherapy delivery are allowed at the discretion of the treating radiation oncologist. This includes continuing a treatment plan which was initiated prior to the start of radiotherapy. A 2-week washout is recommended, but not required.
* Pregnant. Women of childbearing potential must have a negative pregnancy test within 20 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment-related acute toxicity | From start of treatment through 90 days
  -Grade per CTCAE v5.0.
Rate of treatment-related late toxicity | From day 91 through 12 months
  -Grade per CTCAE v5.0.

SECONDARY OUTCOMES:
Change in PRO-CTCAE (General Inventory and Disease Specific Inventory Assessment) | Baseline, at last day of radiotherapy (day 3), within 2 weeks after completion of radiotherapy (day 14), 30 days, 90 days, 180 days, and 360 days
  PRO-CTCAE is a standardized inventory to collected patient reported symptomatic adverse events in clinical trials.
Change in PROMIS Global Health | Baseline, at last day of radiotherapy (day 3), within 2 weeks after completion of radiotherapy (day 14), 30 days, 90 days, 180 days, and 360 days
  PROMIS Global Health is a 10-item patient-reported questionnaire that assesses health related quality of life compared with normal values for the general population with the response options presented as a 5-point (as well as a single 11-point) rating scale. The question that uses an 11-point scale uses a response scale of 0-10 that is recoded to 5 categories (0 = 1; 1-3 = 2; 4-6 = 3; 7-9 = 4; 10 = 5). The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores are indicative of a healthier patient.
Rate of target lesion local control | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Apicelli, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Available data will include de-identified individual participant data collected during the trial.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months after publication. No end date
Access Criteria: Researchers who provide a methodologically sound proposal may be granted data access. Proposals should be directed to apicellia@wustl.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu